CLINICAL TRIAL: NCT01704274
Title: A Double-Blind, Randomised, Placebo-Controlled Study of the Effect of Transdermal Nitroglycerin (Glyceryl Trinitrate; GTN) Therapy on Biomarkers of Immune Escape in Men With Biochemical Recurrence of Prostate Cancer After Primary Therapy
Brief Title: GTN Therapy on Biomarkers of Immune Escape in Men With Biochemical Recurrence of Prostate Cancer After Primary Therapy
Acronym: GTN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. D. Robert Siemens (Other)
Responsible Party: Sponsor-Investigator, Dr. D. Robert Siemens, PI, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Protocol # CAUR 09
Record Dates: First submitted 2012-10-05; First posted 2012-10-11 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: biochemical; recurrence; prostate; cancer; active; surveillence
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence; Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: One arm placebo, two arms different GTN dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo patch
  Interventions: Other: Placebo
- Low dose GTN 0.0285 mg/hr (Experimental): Low dose GTN
  Interventions: Other: Low Dose GTN 0.0285 mg/hr
- High Dose GTN 0.057 mg/hr (Experimental): High Dose GTN
  Interventions: Other: High Dose GTN 0.057 mg/hr

INTERVENTIONS:
Other: Low Dose GTN 0.0285 mg/hr — Low Dose GTN
  Arms: Low dose GTN 0.0285 mg/hr
Other: High Dose GTN 0.057 mg/hr — High Dose GTN
  Arms: High Dose GTN 0.057 mg/hr
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Prostate cancer is the most commonly diagnosed cancer in men in Canada. Over 30% of men over the age of fifty have histological evidence of prostate cancer on biopsy. Despite the stage migration afforded by early detection with serum prostate specific antigen (PSA) testing and an apparent trend toward improved survival over the past several years, prostate cancer remains a significant cause of morbidity and mortality. Biochemical failure after primary therapy (surgery or radiation) remains a significant health care burden and strategies to delay clinical prostate cancer progression and prolong the interval from treatment failure to systemic therapy would be of significant clinical benefit for those men suffering from a finding of PSA recurrence.

PSA is widely accepted as the most useful prognostic marker of prostate cancer progression, particularly after primary therapy with radical surgery or radiation. 5 Despite improved cancer control rates with definitive management of early stage prostate cancer, a PSA recurrence is unfortunately a common occurrence (25-50%) in most large case series.

Microenvironmental factors have been demonstrated to play a pivotal role in the selection of neoplastic cell subpopulations expressing more malignant phenotypes and contributing to the progression of localized and metastatic disease. Very low levels of O2 (< 10 mmHg) has been well described in many solid tumours (including prostate cancer) and the extent of hypoxia has been demonstrated to represent an independent marker of a poor prognosis for patients with various types of cancers. Tumour hypoxia contributes to numerous adaptive phenotypes including increased invasion and metastasis, as well as evasion of immune cell surveillance increased resistance to radiotherapy and chemotherapy. Although cellular adaptive responses to hypoxia are likely mediated by various mechanisms, our previous preclinical studies suggest that decreased nitric oxide (NO)-dependent signalling plays a significant role in this progression of a malignant phenotype.

DETAILED DESCRIPTION:
Researcher's pre-clinical research has demonstrated that hypoxia-induced tumor cell invasiveness, metastatic ability, resistance to chemotherapeutic agents and evasion of immune cell recognition are inhibited by molecules that activate the NO signalling pathway involving cGMP generation (such as glyceryl trinitrate, GTN), and that pharmacological inhibition of NO signalling results in phenotypes similar to those induced by exposure to hypoxia.

Based on pre-clinical data described above the researchers have recently completed and published a phase 2 trial in patients with recurrent prostate cancer using a low-dose, sustained release trasndermal patch of GTN. The GTN was supplied as Minitran™ (nitroglycerin) transdermal delivery system (3M Company, St. Paul, Minnesota) in an open label, non-blinded fashion. GTN is a nitrodonor that has been used in the management of angina for over 100 years with a well-documented safety and tolerability record and has never been associated with carcinogenesis. Their pre-clinical studies have demonstrated that very low molar concentrations of nitric oxide donors are required to attenuate hypoxia-induced malignant phenotypes.

Our results suggest a significant inhibition of progressive disease given the effect on PSA doubling time with GTN treatment compared to their doubling time prior to initiating the trial. Within 12 months of the trial, 17 of 24 patients had doubling times in the slow category or even stable/declining PSA levels. The mean doubling time of the entire cohort increased to 31.8 months from 13.2 months prior to starting treatment. When compared to a matched control group of patients with PSA recurrence that did not receive any treatment, a similar significant difference in PSA doubling time was observed. There were no adverse effects reported in this trial.

This was the first report of the clinical use of nitric oxide donors in the treatment of prostate cancer. The role of nitric oxide in malignant progression has been a subject of controversy, with studies showing either tumor-promoting or tumor-inhibitory roles. These apparently contradictory effects of NO may be explained by the fact that this molecule can regulate phenotypes through a variety of mechanisms depending on local concentrations and the redox state of the cell. Based on our previous findings, the investigators propose that the observed effect of GTN on the PSA of this patient cohort is related to the 'low concentration' effects of NO.

The investigators have identified several possible beneficial mechanisms of effect of low-dose NO donors for cancer management. We have recently published the positive effect of effect of NO signalling (with GTN as the effector molecule) on cancer immune surveillance. The major histocompatibility complex class I chain-related (MIC) molecules, MICA and MICB, play important roles in tumor surveillance by NK cells, lymphokine-activated killer (LAK) cells, and cytotoxic T cells. While MICA is absent from most normal tissues, they can be induced by cellular stresses, such as exposure to carcinogens and infection, and are expressed in a broad range of carcinomas and some haematopoietic malignancies. In humans, the interaction of cell surface MIC molecules with the C-type lectin-like NKG2D receptor on NK, LAK and effector T cells leads to the activation of innate and adaptive immune responses with the subsequent lysis of the tumor cells. Thus, it has been proposed that MIC-NKG2D interactions are critical to the immune surveillance function of NK, LAK and cytotoxic T cells.

The investigators have shown that hypoxia contributes to tumor cell shedding of MIC through a mechanism involving impaired nitric oxide (NO) signalling. While hypoxia increased MIC shedding in human prostate cancer cells, activation of NO signalling inhibited hypoxia-mediated MIC shedding. Similar to incubation in hypoxia, pharmacological inhibition of endogenous NO signalling increased MIC shedding. These findings suggest that the hypoxic tumor microenvironment contributes to impaired immune surveillance and that activation of NO signalling is of potential use in cancer immunotherapy.

Based on previous studies it is investigator's hypothesis that low-dose transdermal GTN will have positive effects on cancer immune surveillance that may translate to therapeutic benefit. In order to establish proof-of-concept, they propose to initiate the correlative study described in this protocol, to determine the effect of the GTN treatment on biomarkers of immune activity in patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males;
* Legal age of consent (18 years of age);
* Histological evidence of adenocarcinoma of the prostate;
* Patients have chosen watchful waiting or active surveillance as preferred management;
* Patients have biochemical failure (defined below) after primary cancer treatment and prefer deferred cancer management:

  * Patients with an increasing PSA at least 3 months after surgery (at least two values above PSA 0.2 ng/mL);
  * Patients with a PSA 2 ng/ml above their nadir PSA after radiation therapy.

Exclusion Criteria:

* Inability to provide an informed consent;
* Inability to adhere to the study protocol for any reason;
* Receiving any other adjuvant therapies for prostate cancer less than 6 months prior to study entry;
* Any contraindication to GTN (including concomitant use of nitroglycerin formulations or phosphodiesterase inhibitors).

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-04; Primary Completion 2017-01 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in the following biomarkers: inflammatory/immune markers uPAR, PAI-1, ULBP2, B7-H1, MIF, TGF-β; and PSA compared to placebo. | 12 months
  All assessments are as per standard of care. The only additional intervention is a 5 mL peripheral vein phlebotomy at each visit. Patients will be followed at 3, 6, 9 and 12 months after initiation of the trial. Clinic visits will assess side effects of drug and include routine follow-up for prostate cancer management. Serum samples for the above-described makers of immune activity will be obtained at the month 3, 6, 9 and 12 visit.

SECONDARY OUTCOMES:
Safety and tolerability of SR low-dose GTN patches in the proposed patient population. | 12 months
  Participant reported safety and tolerability as per FACT-P questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: D. Robert Siemens, MD FRCSC, Principal Investigator — Queen's University
Locations (1):
- Centre for Applied Urological Research/Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided